CLINICAL TRIAL: NCT06609161
Title: A Study to Evaluate the Definitive Bioequivalence of Tedizolid Phosphate Single-Unit-Dose Sachet Powder for Oral Suspension Compared to Tedizolid Phosphate Powder for Oral Suspension Bottle Used in Pediatric Clinical Studies
Brief Title: A Study to Compare Oral Formulations of Tedizolid Phosphate in Healthy Adults (MK-1986-044)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1986-044; MK-1986-044 (Other: MSD)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tedizolid Phosphate Oral Formulation 1 (Reference) (Experimental): Participants will receive oral Formulation 1 (Reference).
  Interventions: Drug: Tedizolid Phosphate Oral Formulation 1 (Reference)
- Tedizolid Phosphate Oral Formulation 2 (Test) (Experimental): Participants will receive oral Formulation 2 (Test).
  Interventions: Drug: Tedizolid Phosphate Oral Formulation 2 (Test)

INTERVENTIONS:
Drug: Tedizolid Phosphate Oral Formulation 1 (Reference) — Formulation 1 (FM1) powder for oral suspension.
  Arms: Tedizolid Phosphate Oral Formulation 1 (Reference)
Drug: Tedizolid Phosphate Oral Formulation 2 (Test) — Formulation 2 (FM2) powder for oral suspension.
  Arms: Tedizolid Phosphate Oral Formulation 2 (Test)

SUMMARY:
The goal of the study is to learn what happens to different oral formulations of tedizolid phosphate (MK-1986) in a healthy person's body over time. Researchers want to know if there is a difference in the oral formulations absorption and elimination from the healthy persons body.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Has body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of or presence of risk factors for Torsades de Pointes (e.g., heart failure/cardiomyopathy or family history of long QT syndrome), or uncorrected hypokalemia or hypomagnesemia
* Has a history of clostridium difficile-associated diarrhea

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the AUC0-Inf of tedizolid.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the AUC0-Last of tedizolid.
Maximum Plasma Concentration (Cmax) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the Cmax of tedizolid.

SECONDARY OUTCOMES:
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 2 weeks postdose
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Number of Participants Who Discontinue Study Drug Due to an AE | Up to approximately 2 weeks postdose
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Time to Maximum Plasma Concentration (Tmax) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the Tmax of tedizolid.
Apparent Terminal Half-Life (t1/2) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the t1/2 of tedizolid.
Apparent Volume of Distribution of Tedizolid During Terminal Phase (Vz/F) | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the Vz/F of tedizolid.
Apparent Clearance (CL/F) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the CL/F of tedizolid.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com